CLINICAL TRIAL: NCT02359526
Title: A Non-randomised, Open-label, Multicenter Phase 4 Pilot Study on the Effect and Safety of Iluvien® in Chronic Diabetic Macular Edema Patients Considered Insufficiently Responsive to Available Therapies With or Without Intravitreal Corticosteroid Therapy (RESPOND)
Brief Title: A Pilot Study on the Effect and Safety of Iluvien® in Chronic Diabetic Macular Edema Patients
Acronym: RESPOND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4C-2014-06
Record Dates: First submitted 2015-02-02; First posted 2015-02-10 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Diabetic Macular Edema
Keywords: Chronic Diabetic Macular Edema; Iluvien; Intra-vitreal injections; Pilot study
MeSH Terms: interventions — Fluocinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ILUVIEN 190 ug intravitreal implant (Experimental): All patients will receive ILUVIEN 190 micrograms intravitreal implant in applicator with an initial release rate of 0.2 microgram per day. The implant will be administered by injection according to the method of administration defined in the SmPC (ILUVIEN SmPC). Only one eye of each patient will be treated with ILUVIEN.
  Interventions: Drug: IlUVIEN

INTERVENTIONS:
Drug: IlUVIEN — All patients will receive ILUVIEN 190 micrograms intravitreal implant in applicator with an initial release rate of 0.2 microgram per day. The implant will be administered by injection according to the method of administration defined in the SmPC (ILUVIEN SmPC). Only one eye of each patient will be treated with ILUVIEN.
  Other Names: Fluocinolone Acetonide

SUMMARY:
To provide treating physicians with experience with ILUVIEN as well as monitoring its safety (and effectiveness) in a real-life chronic diabetic macular edema (DME) patients judged insufficiently responsive to available therapies.

ELIGIBILITY:
Chronic DME patients considered insufficiently responsive to available therapies (laser, anti-VEGF) with or without intravitreal corticosteroid therapy.

Inclusion Criteria:

* Adults (≥18 years) with chronic DME;
* Patients considered as insufficiently responsive as defined as having underwent other previous treatments, including at least 3 anti-VEGF injections in the last 6 months, and the following:

  1. Mean central foveal thickness (central subfield thickness) ≥ 290 um in women and ≥ 305 um in men in Zeiss Cirrus OR ≥ 305 um in women and ≥ 320 um in men in Heidelberg Spectralis, in the study eye as measured using SD-OCT;
  2. Vision impairment (20/50 to 20/400 using Snellen visual acuity equivalent) related to DME;
  3. If in the Investigator's opinion a further improvement is possible.

Exclusion Criteria:

* IOP > 21 mmHg at screening (day -14) in the study eye.
* Historical rise in IOP > 25 mmHg following treatment with an intravitreal corticosteroid in the study eye.
* Use of ≥ 2 active agents as IOP-lowering medications to control IOP at screening in the study eye.
* Vitreomacular traction in DME and opaque media in the study eye.
* Severe proliferative diabetic retinopathy requiring pan retinal photocoagulation in the study eye.
* Pregnant or breastfeeding women.
* Active angiographic central macular ischaemia before baseline in the study eye.
* Pan retinal photocoagulation or cataract surgery 3 months before baseline in the study eye.
* Presence of pre-existing glaucoma, active or suspected ocular or periocular infection and/or hypersensitive to the active agent or to one of the excipients.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant UNLESS they are: using a highly effective method of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Changes in best-corrected visual acuity (BCVA) from baseline to Month-12 | Baseline to 12 months
Changes in central retinal thickness assessed using spectral domain optical coherence tomography (SD-OCT) from baseline to Month-12 | Baseline to 12 months
Occurrence of Adverse events, namely cataract and elevated IOP | 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- Portugal (4):
  - Center for Clinical Trials - Association for Innovation and Biomedical Research on Light and Image, Coimbra
  - Instituto de Retina de Lisboa, Lisbon
  - Hospital de São João, Porto
  - Hospital Vila Franca Xira, Vila Franca de Xira